CLINICAL TRIAL: NCT06379126
Title: The Diagnostic and Prognostic Value of Thrombin-Antithrombin Complex（TAT）, α2-plasmin Inhibitor-plasmin Complex（PIC）, Tissue Plasminogen Activator-inhibitor Complex（tPAI·C） and Thrombomodulin（TM） in Sepsis-induced Coagulopathy
Brief Title: The Diagnostic and Prognostic Value of TAT, PIC, tPAI·C and TM in Sepsis-induced Coagulopathy
Status: Not yet recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: Yuting Li05
Record Dates: First submitted 2024-04-17; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Sepsis-induced Coagulopathy
Keywords: sepsis-induced coagulopathy; biomarker; diagnostic value

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SIC group: SIC score≥4
  Interventions: Diagnostic Test: Test thrombin-antithrombin complex（TAT）, α2-plasmin inhibitor-plasmin complex（PIC）, tissue plasminogen activator-inhibitor complex（tPAI·C） and thrombomodulin（TM）
- non-SIC group: SIC score<4
  Interventions: Diagnostic Test: Test thrombin-antithrombin complex（TAT）, α2-plasmin inhibitor-plasmin complex（PIC）, tissue plasminogen activator-inhibitor complex（tPAI·C） and thrombomodulin（TM）

INTERVENTIONS:
Diagnostic Test: Test thrombin-antithrombin complex（TAT）, α2-plasmin inhibitor-plasmin complex（PIC）, tissue plasminogen activator-inhibitor complex（tPAI·C） and thrombomodulin（TM） — Test TAT, PIC, tPAI·C and TM of blood of SIC patients.

SUMMARY:
In order to evaluate the diagnostic and prognostic value of thrombin-antithrombin complex（TAT）, α2-plasmin inhibitor-plasmin complex（PIC）, tissue plasminogen activator-inhibitor complex（tPAI·C） and thrombomodulin（TM） in sepsis-induced coagulopathy(SIC), hospitalized patients with sepsis were prospectively included. Plasma TAT, PIC, tPAI·C,TM levels within 24 h after sepsis diagnosis were detected by MCL60 chemiluminescence analyzer. According to the SIC score (≥4), they were divided into SIC group and non-SIC group, and ROC curve analysis was performed according to the biomarker test results.

DETAILED DESCRIPTION:
Thrombin-antithrombin complex（TAT）, α2-plasmin inhibitor-plasmin complex（PIC）, tissue plasminogen activator-inhibitor complex（tPAI·C） and thrombomodulin（TM） can evaluate vascular endothelial damage, thrombin and plasminase activation, and have clinical significance in early diagnosis of DIC, thrombotic disease and monitoring of thrombolysis efficacy. However, whether these biomarkers can be used for early diagnosis of SIC is unclear.

In order to evaluate the diagnostic value of TAT, PIC, tPAI·C and TM in sepsis-induced coagulopathy(SIC), hospitalized patients with sepsis were prospectively included. Plasma TAT, PIC, tPAI·C,TM levels within 24 h after sepsis diagnosis were detected by MCL60 chemiluminescence analyzer. According to the SIC score (≥4), they were divided into SIC group and non-SIC group, and receiver operator characteristic（ROC） curve analysis was performed according to the biomarker test results. The area under the curve(AUC) was used to determine whether TAT, PIC, tPAI·C and TM could be used as biomarkers for SIC diagnosis. If AUC is between 0.7 and 0.9, this indicator has diagnostic value.

ELIGIBILITY:
Inclusion Criteria:

* Septic patients who meet the diagnostic criteria of sepsis 3.0.

Exclusion Criteria:

* age < 18 years old, heparin induced thrombocytopenia, thrombotic thrombocytopenic purpura, antiphospholipid syndrome or liver cirrhosis classified as Child-Pugh grade C and patients with a current treatment that interfered with coagulation (anticoagulants).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Septic patients who meet the diagnostic criteria of sepsis 3.0 admitted to the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Thrombin-antithrombin complex（TAT）, α2-plasmin inhibitor-plasmin complex（PIC）, tissue plasminogen activator-inhibitor complex（tPAI·C） and thrombomodulin（TM） level | 4 hours
  Plasma TAT, PIC, tPAI·C,TM levels within 24 h after sepsis diagnosis were detected by MCL60 chemiluminescence analyzer. According to the SIC score (≥4), they were divided into SIC group and non-SIC group, and receiver operator characteristic （ROC）curve analysis was performed according to the biomarker test results. The area under the curve(AUC) was used to determine whether TAT, PIC, tPAI·C and TM could be used as biomarkers for SIC diagnosis. If AUC is between 0.7 and 0.9, this indicator has diagnostic value.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Zhang, Study Director — The First Hospital of Jilin University

IPD SHARING:
Plan to Share IPD: No